CLINICAL TRIAL: NCT03264586
Title: The Effect of Lidocaine - Prilocaine Cream (EMLA) Versus Mepivacaine Infiltration on Pain Relief During And After Mediolateral Episiotomies: A Randomized Clinical Trial
Brief Title: The Effect of Lidocaine - Prilocaine Cream (EMLA) Versus Mepivacaine Infiltration on Pain Relief During And After Mediolateral Episiotomies
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 9
Record Dates: First submitted 2017-08-25; First posted 2017-08-29 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Episiotomy Pain
MeSH Terms: interventions — Lidocaine, Prilocaine Drug Combination; Mepivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine-prilocaine cream (Active Comparator): Women who were assigned randomly to receive EMLA cream had a 5gm dose of cream applied to the intact surface of the perineum and area covered with an occlusive dressing to facilitate pemetration thrug stratum corneum
  * EMLA cream was applied, 1 hour before the expected time of birth.
  * With the assistance at birth, the residue of cream was removed to prevent contact with the fetus, because sodium hydroxide, which is a component of the cream, can cause fetal eye irritation.
  * No additional anesthetic was applied if episiotomy was necessary.
  * Before commancement of perineal repair any residual cream was wiped off.
  Interventions: Drug: Lidocaine-prilocaine cream; Procedure: mediolateral episiotomy
- mepivacaine infiltration group (Active Comparator): * In the mepivacaine group, 10 ml of 1% mepivacaine solution was injected slowly when the fetal head was crowned with frequent aspiration to avoid intravascular injection.
  * In the mepivacaine group, if an episiotomy was indicated, it was performed after infiltration of perineal tissue with 10 ml of 1% mepivacaine solution.
  * The suture procedure was delayed 10 minutes after the injection of the aneathetic
  Interventions: Drug: mepivacaine infiltration group; Procedure: mediolateral episiotomy

INTERVENTIONS:
Drug: Lidocaine-prilocaine cream — 5gm dose of cream applied to the intact surface of the perineum and area covered with an occlusive dressing to facilitate penetration
  - EMLA cream was applied, 1 hour before the expected time of birth.
  Other Names: EMLA cream
  Arms: Lidocaine-prilocaine cream
Drug: mepivacaine infiltration group — 10 ml of 1% mepivacaine solution was injected slowly when the fetal head was crowned with frequent aspiration to avoid intravascular injection.
  * In the mepivacaine group, if an episiotomy was indicated, it was performed after infiltration of perineal tissue with 10 ml of 1% mepivacaine solution.
  * The suture procedure was delayed 10 minutes after the injection of the aneathetic
  Other Names: 1% mepivacaine
  Arms: mepivacaine infiltration group
Procedure: mediolateral episiotomy — Episiotomy repair a loose, continous, non locking suture to close the vaginal mucosa and the muscular layer of the perineum using vicryl Number zero (0).
  * At the end of the vaginal mucosal repair care is taken to align the edges of the episiotomy wound
  * At the point where perineal skin begins; the suture is then passed beneath the vaginal mucosa, and repair of perineal muscle begins. The deep layer of muscles is closed first, ensuring no dead space one left behind
  * The skin was closed with the same continuous suture to approximate the subcutinuous tissue.

SUMMARY:
Included women were divided randomly into two groups:

Group A: (n=100): women were subjected to application of EMLA® cream "Lidocaine-prilocaine cream (EMLAcream; Astra Zeneca, Basiglio, Italy is an entectic mixture of 2.5% lidocaine and 2.5% prilocaine)"for pain relief during episiotomy repair.

Group B: (n=100): women were subjected to application of local injection of 10 ml of 1% mepivacaine for pain relief during episiotomy repair.

DETAILED DESCRIPTION:
During the second stage of labor, women were placed in the lithotomy position. 10- Patients who were enrolled in the study were guaranteed to obtain additional anesthesia during episiotomy repair whenever pain exceeded the tolerability threshold.

11- Volunteers were assigned randomly to have either local injection of 10 ml of 1% mepivacaine or application of 5gm-dose® EMLA cream"Lidocaine- prilocaine cream(EMLA cream; Astra Zeneca, Basiglio, Italy is an entectic mixture of 2.5% lidocaine and 2.5% prilocaine)" for pain relief during episiotomy repair.

1. Group A: "EMLA group"

   * Women who were assigned randomly to receive EMLA cream had a 5gm dose of cream applied to the intact surface of the perineum and area covered with an occlusive dressing to facilitate pemetration thrug stratum corneum
   * EMLA cream was applied, 1 hour before the expected time of birth.
   * With the assistance at birth, the residue of cream was removed to prevent contact with the fetus, because sodium hydroxide, which is a component of the cream, can cause fetal eye irritation.
   * No additional anesthetic was applied if episiotomy was necessary.
   * Before commancement of perineal repair any residual cream was wiped off.
2. Group B: "mepivacaine infiltration group".

   * In the mepivacaine group, 10 ml of 1% mepivacaine solution was injected slowly when the fetal head was crowned with frequent aspiration to avoid intravascular injection.
   * In the mepivacaine group, if an episiotomy was indicated, it was performed after infiltration of perineal tissue with 10 ml of 1% mepivacaine solution.
   * The suture procedure was delayed 10 minutes after the injection of the aneathetic
   * All episiotomies were performed at the top of contraction as mediolateral episiotomies.

     12- Episiotomy repair
   * In all cases episiotomies was repaired with a loose, continous, non locking suture to close the vaginal mucosa and the muscular layer of the perineum using vicryl Number zero (0).
   * The suture begins about 0.5 cms above the apex of the vaginal wound The suture are evenly placed to allow for approximation of the edges of the wound without causing tension or wrinkling or over lapping.
   * At the end of the vaginal mucosal repair care is taken to align the edges of the episiotomy wound to restore the appearance of the hymenal ring, the fourchette and the beginning of the perineal skin.
   * At the point where perineal skin begins; the suture is then passed beneath the vaginal mucosa, and repair of perineal muscle begins. The deep layer of muscles is closed first, ensuring no dead space one left behind, and ensuring no bleeding points are ignored.
   * The skin was closed with the same continuous suture to approximate the subcutinuous tissue.
   * The wound is cleared with antiseptic solution and covered by addressing. 14- Before leaving the delivery suite (approximately 2 hours after delivery) each patient was asked to record the severity of pain that she had experienced during perineal repair in a 10-cm visual analog scale, where 0 cm means no pain and 10 cm means unbearable pain.
   * The patient was asked to mark the point that best indicated the perception of her pain on the visual analog scale
   * Finally, women were asked to express their overall satisfaction with the anesthesia method during perineal repair with "yes" or "no" answers

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age 37 weeks or more
2. Singleton gestation.
3. Uncomplicated pregnancy.
4. Vertex presentation.

Exclusion Criteria:

1. Epidural analgesia request.
2. Operative delivery.
3. No other methods are used for pain control 2hours befor episiotomy
4. Previous adverse reaction to local anesthetic.

Ages: 19 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
pain | 24 hours after delivery
  The patient was asked to mark the point that best indicated the perception of her pain on the visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — kasr Alainy medical school
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt